CLINICAL TRIAL: NCT04509193
Title: RIVA-DM: Effectiveness and Safety of Rivaroxaban vs. Warfarin in Nonvalvular Atrial Fibrillation and Diabetes Mellitus: Analysis of Electronic Health Record Data
Brief Title: A Study Using Electronic Health Information to Learn About Rivaroxaban Compared to Warfarin in Participants With Non-valvular Atrial Fibrillation (NVAF) and Diabetes
Acronym: RIVA-DM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 21449; EUPAS36634 (Other: ENCePP)
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants with diagnoses of type 2 diabetes and non-valvular atrial fibrillation (NVAF) newly-initiated on rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Group B: Participants with diagnoses of type 2 diabetes and non-valvular atrial fibrillation (NVAF) newly-initiated on warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Participants receive rivaroxaban (per written prescription, medication administration or self-report of medication use)
  Groups: Group A
Drug: Warfarin — Participants receive warfarin (per written prescription, medication administration or self-report of medication use)
  Groups: Group B

SUMMARY:
In people with type 2 diabetes, the body does not make enough of a hormone called insulin or does not use insulin well. This results in high blood sugar levels.

People with diabetes are more likely to have non-valvular atrial fibrillation (NVAF) compared to people who do not have diabetes. Having both NVAF and diabetes can increase the chances of developing other serious health conditions, like blood clots and strokes.

People with NVAF may receive treatments to help lower the risk of blood clots. This can then help to lower the risk of having a stroke. Two of these treatments are rivaroxaban and warfarin.

In this study, the researchers will look at how well rivaroxaban works and how safe it is compared to warfarin in routine clinical practice. The study will include men and women who are at least age 18 and who have NVAF and type 2 diabetes.

The researchers in this study will use the participants' health information from an electronic database.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age at the time of anticoagulation initiation
* Have diagnoses of type 2 diabetes and Non-valvular atrial fibrillation (NVAF)
* Have no record of prior oral anticoagulant (OAC) use in the prior 12-months
* Newly initiated on Rivaroxaban or Warfarin (index date)
* Have ≥12-months of electronic health record (EHR) activity prior to the index date and received care documented in the EHR database from at least one provider in the 12-months prior

Exclusion Criteria:

* Evidence of valvular heart disease defined as any rheumatic heart disease, mitral stenosis or mitral valve repair/replacement
* Pregnancy
* Use of rivaroxaban doses other than 15 mg once daily or 20 mg once daily or the presence of other indication(s) for OAC use
* Any prior OAC utilization per written prescription or self-report at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is using Optum electronic health record (EHR) database. The study population of interest will be US participants with Non-valvular atrial fibrillation (NVAF) and comorbid type 2 diabetes, oral anticoagulation (OAC)-naïve and newly-initiated on rivaroxaban or warfarin, be active in the data set and have received care.
Sampling Method: Non-Probability Sample
Enrollment: 116049 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Composite of stroke or systemic embolism | Up to 8 years
Any major or clinically-relevant nonmajor bleed resulting in hospitalization | Up to 8 years

SECONDARY OUTCOMES:
Ischemic stroke | Up to 8 years
Systemic embolism | Up to 8 years
Need for revascularization or major amputation of the lower limb | Up to 8 years
Intracranial hemorrhage | Up to 8 years
Critical organ bleeding per ISTH categories | Up to 8 years
  The categories for critical organ bleeding as per ISTH definition are: intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome.
Any extracranial bleeding | Up to 8 years
Any hospitalization due to intracranial or critical organ bleeding or a bleed in another location associated with either a 2 g/dL drop in hemoglobin or need for transfusion | Up to 8 years
Doubling of the serum creatinine level from baseline | Up to 8 years
Decrease in eGFR>30% or 40% | Up to 8 years
  Glomerular filtration rate (GRF)
Development of an eGFR<15 mL/min or initiation of dialysis | Up to 8 years
  Glomerular filtration rate (GRF)
Development of end-stage renal disease per billing codes only | Up to 8 years
Development of urine albumin-to-creatinine ratio (UACR) of 30-300 or >300 | Up to 8 years
Development of serum potassium > 5.6 or >6 mg/dL | Up to 8 years
Development of diabetic retinopathy | Up to 8 years
Myocardial infarction | Up to 8 years
All-cause mortality | Up to 8 years
Vascular mortality | Up to 8 years
Major adverse cardiovascular event | Up to 8 years
Composite of stroke, systemic embolism, vascular death | Up to 8 years
Composite of stroke, systemic embolism, myocardial infarction, vascular death | Up to 8 years
Composite stroke, systemic embolism, need for lower limb revascularization or major amputation | Up to 8 years
Composite of >40% decrease in eGFR from baseline, eGFR<15 mL/minute, need for dialysis, renal transplant, major adverse limb event, retinopathy or all-cause death | Up to 8 years
  Glomerular filtration rate (GRF)
New-onset vascular dementia | Up to 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- US Optum De-Identified EHR data, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Costa OS, O'Donnell B, Vardar B, Abdelgawwad K, Brescia CW, Sood N, Coleman CI. Kidney, limb and ophthalmic complications, and death in patients with nonvalvular atrial fibrillation and type 2 diabetes prescribed rivaroxaban or warfarin: an electronic health record analysis. Curr Med Res Opin. 2021 Sep;37(9):1493-1500. doi: 10.1080/03007995.2021.1947217. Epub 2021 Jul 8. PMID 34166150
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/